**Document Date:** April 7, 2020

EFFECT OF EXPIRATORY MUSCLE TRAINING ON STOMATOGNATHIC

SYSTEM IN PATIENTS WITH STROKE

Ömer DURSUN PT, PhD<sup>1</sup>. Tamer ÇANKAYA, PT, Assoc. Prof. Dr<sup>2</sup>. Erdal DİLEKÇİ, MD, Assoc. Prof. Dr<sup>3</sup>.

STUDY PROTOCOL

The aim of this study was to analyze and assess the effect of expiratory muscle training

on the stomatognathic system in patients with stroke. Total of 31 individual included as 16

control and 15 study group to the study. Temporomandibular joint range of motion,

masticatory muscle pressure pain threshold, facial asymmetry existence, head posture, oral

hygiene health and habit, masticatory performance, intraoral pH, deglutition function and

deep neck flexor muscle endurance of the individuals was assessed in order by; digital

caliper, algometry, labial commissure and craniocervical angle measurement, general oral

health assessment index and questionnaire, sieve test, digital pH gauge, repetitive saliva

swallow test and, eating assessment tool and deep neck flexor endurance test. While study

group was enrolled to 3-week respiratory muscle training in addition to conventional

physiotherapy, control group enrolled to the conventional physiotherapy programme.

NCT NUMBER: NCT04569968